CLINICAL TRIAL: NCT02565303
Title: Minimum Effective Dose of Intrathecal Ropivacaine Required for Cesarean Delivery: A Prospective, Randomized Comparison Between L2-3 and L3-4 Approach
Brief Title: Minimum Effective Dose of Ropivacaine for Spinal Anesthesia for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng WANG, physician, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-35-(1)
Record Dates: First submitted 2015-09-19; First posted 2015-10-01 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Spinal Anesthesia
Keywords: cesarean delivery; ropivacaine; minimum effective dose; dose-response relationship; intrathecal; intervertebral space
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L2-3 intervertebral group (Experimental): The initial dose of ropivacaine for subarachnoid is chosen as 12 mg in L2-3 intervertebral space group.
  Interventions: Procedure: Intervertebral space; Drug: Ropivacaine
- L3-4 intervertebral group (Experimental): The initial dose of ropivacaine for subarachnoid is chosen as 15 mg in L3-4 group.
  Interventions: Procedure: Intervertebral space; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Intervertebral space
Drug: Ropivacaine — The initial dose of ropivacaine is chosen as 12 mg in L2-3 group and 15 mg in L3-4 group with the volume of 3 mL in both groups. The testing interval is 0.5 mg with subsequent doses being determined by the outcome of the previous injection in the same group.If the previous response is ineffective, the next patient will receive 0.5 mg more than the last patient. If the response of the previous patient is effective, the next patient decrease 0.5mg.
  Other Names: Naropin

SUMMARY:
Ropivacaine is one of commonly used anesthetics for spinal anesthesia. Usually L2-3 or L3-4 intervertebral space is chosen for spinal anesthesia. The efficacy of ropivacaine injected into subarachnoid space depends on the given dose and the chosen intervertebral space. Appropriate dose could satisfy the requirement of operation and reduce incidence of the adverse reaction. But it is not certain about the minimum effective dose of ropivacaine in cesarean section through the two intervertebral spaces, respectively. This study is being conducted to find the minimum effective doses for L2-3 and L3-4 spinal anesthesia in cesarean section.

DETAILED DESCRIPTION:
Some unexpected adverse reactions such as respiratory depression, vomiting, especially supine hypotensive syndrome could caused by a high dose of anesthetic in cesarean section. The investigators assumed that there be a minimum effective dose that will be associated with the best possible performance of ropivacaine for different intervertebral spaces(L2-3 and L3-4 in usual). That maybe enhance the comfort of parturient and safety of fetus.

This study is conducted as a prospective, randomized, up-down sequential dose of isobaric ropivacaine in 3 mL that will provide effective analgesia for 50% of parturients in cesarean section. The investigators use the combined spinal-epidural anesthesia(CSEA) technique in the study. The initial dose of ropivacaine is chosen as 12 mg in L2-3 group and 15 mg in L3-4 group, and the testing interval is 0.5 mg with subsequent doses being determined by the outcome of the previous injection in the same group. If the previous response is ineffective, the next patient will receive 0.5 mg more than the last patient. If the response of the previous patient is effective, the next patient decrease 0.5mg.

The visual analogue scale (VAS) is used to rate the pain, where 0 is no pain and 10 is the worst pain imaginable. Criteria for evaluation:(1) effective: after spinal anesthesia finish, a dose that provide adequate sensory dermatomal anesthesia to pinprick to T6 or higher within 10 minutes, and the VAS is lower than or equal to 3 within 60minutes after skin incision; (2) ineffective: if the initial plane of sensory dermatomal anesthesia is lower than T6 or VAS is greater than 3 within 60 minutes after skin incision, the dose of ropivacaine is considered inadequate and additional lidocaine is given through epidural catheter.

Motor assessments are performed at the start of operation. Motor block in the lower limb is assessed by a modified Bromage scale (0=no paralysis, 1=unable to raise extended leg, 2=unable to flex knee,3=unable to flex ankle). All of the assessments are made by an anesthetist who is blinded to the group assignment as well as to the dose injected.

On the other hand, the investigators will compare the incidence of adverse reaction between the L2-3 and L3-4 group.

Using the Dixon and Massey up-and-down method study design, 60 patients scheduled for elective cesarean section will be included in the study, 30 for each group.

ELIGIBILITY:
Inclusion Criteria:

* Full term parturient(> 37 and <42 weeks gestation)
* Above 20 years and below 35 years
* American Society of Anesthetists(ASA) I to II
* Singleton pregnancy
* Elective cesarean section
* Body weight during 60-85kg, height during 150-170cm

Exclusion Criteria:

* Patient refusal
* Hypertension
* Diabetes mellitus
* Heart diseases
* Asthma
* Abnormal fetus or placenta
* Contraindications to combined spinal-epidural anesthesia(CSEA)
* Allergy to ropivacaine

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
sensory block assessment evaluated with visual analogue scale (VAS) and sensory dermatomal anesthesia | during the entire procedure of operation
  Sensory block assessment will be evaluated with VAS and sensory dermatomal anesthesia. Criteria for evaluation of anesthetic efficacy:(1) effective: within 10 minutes after intrathecal injection, a dose that provides adequate sensory dermatomal anesthesia to pinprick to T6 or higher, and the VAS is lower than or equal to 3 within 60minutes after skin incision; (2) ineffective: the initial plane of sensory dermatomal anesthesia is lower than T6 or VAS is higher than 3 within 60 minutes after skin incision. VAS is a psychometric response scale which can be used in questionnaires. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points, where 0 was no pain and 10 was the worst. A dermatome is an area of skin that is mainly supplied by a single spinal nerve.Usually the upper sensory dermatomal anesthesia is used to assess the effect of intrathecal anesthesia.

SECONDARY OUTCOMES:
motor block accessment | 10minutes after the spinal anesthesia finished
  Motor block in the lower limb will be assessed by a modified Bromage scale (0=no paralysis, 1=unable to raise extended leg, 2=unable to flex knee,3=unable to flex ankle) .

OTHER OUTCOMES:
incidence of adverse reaction | during the entire procedure of operation
  The investigators will compare the incidence of adverse reaction between the L2-3 and L3-4 group such as maternal hypotension, bradycardia, respiratory depression, nausea and vomiting.
effect of abdominal muscle relaxation | during the entire procedure of operation
  The quality of abdominal muscle relaxation will be evaluated by the obstetrician as excellent (no disturbing muscle strain), satisfactory (disturbing, but acceptable) or unsatisfactory (unacceptable).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China